CLINICAL TRIAL: NCT05793307
Title: A Multi-centered, Single Arm, Open Labeled, Study to Evaluate the Safety and Efficacy of an Adeno-associated Virus Vector Expressing the Human Acid Alpha-glucosidase (GAA) Transgene Intravenous Injection in Patients With Infantile-onset Pompe Disease
Brief Title: Evaluation of the Safety and Efficacy of Infantile-onset Pompe Disease Gene Therapy Drug
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC301-IOPD-001
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pompe Disease Infantile-Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Single intravenous administration of GC301 at a dose of 8.0 x 10^13 vector genomes per kilogram body weight
  Interventions: Genetic: GC301
- Cohort 2 (Experimental): Single intravenous administration of GC301 at a dose of 1.2 x 10^14 vector genomes per kilogram body weight
  Interventions: Genetic: GC301
- Cohort 3 (Experimental): Single intravenous administration of GC301 at a dose of 1.8 x 10^14 vector genomes per kilogram body weight
  Interventions: Genetic: GC301

INTERVENTIONS:
Genetic: GC301 — GC301, is an adeno-associated virus 9 (AAV9) vector delivering a functional copy of the human GAA gene

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of GC301 adeno-associated virus vector expressing codon-optimized human acid alpha-glucosidase (GAA) as potential gene therapy for Pompe disease. Patients diagnosed with infantile-onset Pompe disease who are younger than 6 months old will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age < 6 months
* Patient has diagnosis of infantile onset Pompe disease
* The patient's legal guardian(s) must be able to understand the purpose and risks of the study and voluntarily provide signed and dated informed consent prior to any study-related procedures being performed.

Exclusion Criteria:

* Left ventricle ejection fraction (LVEF) < 40%;
* Patient who has AAV9 neutralizing antibody titer ≥ 1:100；
* Patient who has received enzyme replacement therapy (ERT) more than twice;
* Patient who has respiratory dysfunction before enrollment, including the blood oxygen (O2) saturation level < 90%, or the partial pressure of carbon dioxide (PCO2) in venous blood > 55 mmHg, or PCO2 in arterial blood > 40 mmHg;
* Patient who has laboratory abnormalities of: creatinine > Upper Limit of Normal (ULN), hemoglobin < 90 g/L;
* Patient with congenital organ absence;
* Patient with a history of glucocorticoid allergy;
* Patient who is positive for human immunodeficiency (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or treponema pallidum antibody;
* Patient who has participated in a previous gene therapy research trial;
* Patient who has any concurrent clinically significant major disease or any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in the study.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability over time | 52 weeks
  Frequency of adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests
Proportion of patients treated with GC301 who are alive | 52 weeks

SECONDARY OUTCOMES:
Proportion of patients treated w/ GC301 who were alive and free of ventilator support | 52 weeks
Changes from baseline Left Ventricular Mass (LVM) annd LVMI (LVM index) | 26 and 52 weeks
Changes from baseline creatine kinase (CK), CK-MB, Troponin I, B-Type Natriuretic Peptide (BNP) | 26 and 52 weeks

OTHER OUTCOMES:
Change from baseline glycogen content in muscle tissue | 26 and 52 weeks
Change from baseline acid alpha-glucosidase (GAA) enzyme in muscle and blood | 26 and 52 weeks
Change in patient's motor function | 52 weeks
  To evaluate the changes in patient's mobility and physical ability using Hammersmith Infant Neurological Examination (HINE) scores
The viral load of adeno-associated virus (AAV) vector | At multiple time points from pre-dose through up to 1 years post-dose
  To assess the change of AAV vector copy numbers within 52 weeks after administration.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking Union Medical College, Beijing
  - 301 Chinese PLA General Hospital, Beijing
  - Central South University, Xiangya Hospital, Changsha
  - Zhejiang University, School of Medicine, The Children's Hospital, Hangzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou